CLINICAL TRIAL: NCT00503620
Title: The Effect of Botulinum Toxin on Neuromuscular Function in the Child With Cerebral Palsy
Brief Title: The Effect of Botox on Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: United Cerebral Palsy Foundation (Other)
Responsible Party: Richard T. Lauer, Shriners Hospitals for Children
Other Study IDs: R-784-06
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Botulinum Toxin; Neuromuscular Function
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum Toxin A — Injection into the gastrocnemius/soleus muscles for spasticity

SUMMARY:
Botulinum toxin injections are a common form of treatment for children with cerebral palsy to help reduce muscle tightness and help them walk without resorting to surgery. While the treatment is beneficial, it requires that the therapy be repeated every six months, which can be costly and may eventually result in the therapy not being effective over time. The study being conducted at Shriners Hospitals for Children, Philadelphia, will examine the effects of botulinum toxin injections, not only on walking, but on the changes it causes in the muscle, brain and spinal cord. The changes in the muscle, brain and spinal cord, called neuromuscular plasticity, have not been extensively examined in response to botulinum toxin, and could provide insight into how botulinum toxin works and how to make it more effective. This study will focus on children with cerebral palsy between the ages of 4 and 12 years, with only one leg involved and who would normally be receiving botulinum toxin injections of the lower leg to help improve walking. The children will be asked to come into the hospital for a full day before they receive the injection, and then again after four and twelve weeks to look at the changes in the muscle, brain and spinal cord. This will involve recording them while they walk, measurements of the muscle reflexes, and recording their brain activity while the move their ankle (also known as functional magnetic resonance imaging or fMRI). A group of children with typical development will also be asked to participate in the study to act as a comparison group. The researchers believe that examining the changes in the muscles, brain and spinal cord in response to the injection will aid in the understanding how better to use botulinum toxin to achieve better or longer lasting changes.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of spastic hemiplegic or diplegic CP
2. Children must be ambulatory without the use of assistive devices
3. Children must be between the ages of 4 and 12 years
4. Children must be cleared by an orthopedic surgeon for risk of hip subluxation or dislocation and cannot have significant scoliosis (curvature > 40 degrees)
5. Children must be seizure-free or seizure controlled
6. Children must have visuoperceptual skills and cognitive/communication skills sufficient to follow multiple step commands and to attend to tasks associated with data collection
7. Children's passive range of motion in lower extremity joints must be less than 20 degrees of flexion contracture at the hips as measured by the Thomas Test, at least 20 degrees of hip abduction bilaterally, les than 0 degrees of knee flexion contracture, popliteal angle less than 55 degrees, and at least 0 degrees of ankle dorsiflexion with the knee extended while the foot is in varus
8. Children who are planning to undergo botulinum toxin injections of the gastrocnemius and/or soleus muscles without serial casting as clinically dictated for the treatment of muscle spasticity

Exclusion Criteria:

1. Children who have a diagnosis of "mixed" types of CP (i.e. athetosis) or other movement disorders (i.e. ataxia)
2. Children who have had a selective dorsal rhizotomy, are presently are receiving intrathecal Baclofen, or have changed their spasticity medications in the past 6 months.
3. Children who have a metallic or electrical implants
4. Children who are unable to stay in the MRI machine for the 8 to 10 minute duration of the exam.
5. Children who have a history of claustrophobia.
6. Female children cannot be pregnant. A pregnancy test will be given if it is possible that the child can become pregnant, to ascertain whether or not the child is pregnant.
7. Children who are planning to receive serial casting post botox injection.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic hemiplegic or diplegic CP, GMFCS Level I or II
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-01; Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lauer, PhD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Philadelphia, Pennsylvania, United States